CLINICAL TRIAL: NCT04631016
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety and Tolerability of MEDI3506 in Participants With Moderate to Severe Chronic Obstructive Pulmonary Disease and Chronic Bronchitis (FRONTIER 4)
Brief Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Assess MEDI3506 in Participants With COPD and Chronic Bronchitis
Acronym: FRONTIER-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9180C00002; 2020-000571-20 (EudraCT Number)
Record Dates: First submitted 2020-10-20; First posted 2020-11-16 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Chronic Bronchitis
Keywords: MEDI3506; IL-33; COPD; Chronic Bronchitis; Lung function; Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to recieve either MEDI3506 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational product only will be prepared and administrated by unmasked personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tozorakimab (Experimental): Participants received 7 doses of subcutaneous (SC) tozorakimab Dose Level 1 injection once every 4 weeks (Q4W).
  Interventions: Drug: Tozorakimab
- Placebo (Placebo Comparator): Participants received 7 doses of SC placebo injection matched to tozorakimab once Q4W.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tozorakimab — Participants will receive SC injection of tozorakimab as stated in arm description.
  Other Names: MEDI3506
  Arms: Tozorakimab
Other: Placebo — Participants will receive SC injection of placebo as stated in arm description.
  Arms: Placebo

SUMMARY:
This is a research study to determine the efficacy and safety of investigational drug MEDI3506 for the treatment of adult participants with Chronic Obstructive Pulmonary Disease and Chronic Bronchitis.

DETAILED DESCRIPTION:
Study D9180C00002 is a Phase II, randomised, double-blind, placebo-controlled, parallel group, proof of concept study to evaluate the efficacy and safety of MEDI3506 in adult participants with moderate to severe Chronic Obstructive Pulmonary Disease and Chronic Bronchitis.

Approximately 85 sites globally will participate in this study. Approximately 144 participants will be randomized to 2 treatment groups in a 1:1 ratio to receive MEDI3506 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Participant must be 40 to 80 years of age inclusive, at the time of signing the informed consent form (ICF).
* Participants who are current or ex-smokers with a tobacco history of >= 10 pack-years.
* Participants who have a documented history of COPD for at least 1 year.
* Participants who have a post-BD FEV1/FVC < 0.70 and a post-BD FEV1 >= 20% and < 80% predicted normal value at screening. Centralized spirometry will be used for this criteria assessment.
* Participants who have a physician confirmed participant history of chronic bronchitis as defined as presence of cough and sputum on most days for >= 3 months/year in at least the 2 year period immediately prior to study visit 1 (SV1) (Screening).
* Participants who have an average BCSS score of >= 2 in cough and >= 2 in sputum domains assessed over 14 days preceding SV3.
* Participants who have a documented stable regimen of dual therapy or triple therapy for >= 3 months prior to enrolment; there should have been no change in treatment after the previous exacerbation prior to entering into the study. Where dual therapy consists of inhaled corticosteroids (ICS) + long-acting beta 2 agonist (LABA) or LABA + long-acting muscarinic receptor antagonist (LAMA), and triple therapy consists of ICS + LABA + LAMA.
* Participants who have a documented history of >= 1 moderate or severe AECOPD requiring systemic corticosteroids and/or antibiotics for at least 3 days duration (or 1 injection of depot formulation), or hospitalization for reason of AECOPD in the previous 24 months.
* Body mass index within the range 18 to 40 kg/m^2 (inclusive).
* Female participants of childbearing potential, must have negative pregnancy tests.
* Male and female participants must follow protocol contraceptive guidance.

Exclusion Criteria:

* Participants with a positive diagnostic nucleic acid test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at screening. Participants with mild or asymptomatic disease could be rescreened.
* Participants with a significant coronavirus disease 2019 (COVID-19) illness within 6 months of enrolment.
* As judged by the investigator, any evidence of any active medical or psychiatric condition or other reason which in the investigator's opinion makes it undesirable for the participant to participate in the study.
* Current or past diagnosis of asthma which persisted beyond age of 25 years.
* Clinically important pulmonary disease other than COPD, radiological findings, and/or laboratory findings suggestive of a respiratory disease other than COPD that is contributing to the participant's respiratory symptoms.
* Increased pre-BD FEV1 at randomization visit (SV3) compared to Screening SV1 of >= 400 mL or >= 25% of SV1 FEV1.
* Any other clinically relevant abnormal findings on physical examination, laboratory testing; or chest CT scan, which in the opinion of the investigator or medical monitor may compromise the safety of the participant in the study or interfere with evaluation of the study intervention or reduce the participant's ability to participate in the study.

Chest CT scan findings requiring further investigation or repeat CT surveillance before SV14.

* A family history of heart failure.
* A LVEF < 45% measured by echocardiogram.
* History of a clinically significant infection (viral, bacterial, or fungal) within 4 weeks.
* History of, or a reason to believe a participant has a history of, drug or alcohol abuse within the past 2 years prior to screening.
* Participants with a recent history of, or who have a positive test for, infective hepatitis or unexplained jaundice, or participants who have been treated for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Evidence of active or untreated latent tuberculosis (TB).
* Change in smoking status in 12 weeks prior to enrolment or intention to change smoking status between enrolment and end of follow-up.
* Participants currently receiving background therapy that is not approved by regulatory authorities in the country of study for COPD are not eligible for the study.
* History of treatment with cardiotoxic medications (eg, as part of cancer therapy) including thiazolidinedione's.
* Treatment with broad spectrum antibiotic within 4 weeks prior to randomization (Day 1).
* Receiving any of the prohibited concomitant medications as specified in the clinical study protocol (CSP).
* Inability to perform technically acceptable spirometry.

Additional inclusion and exclusion criteria's applies.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (85):
- United States (16):
  - Research Site, Sheffield, Alabama
  - Research Site, Newport Beach, California
  - Research Site, Newark, Delaware
  - Research Site, Kissimmee, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Lakeside Park, Kentucky
  - Research Site, White Marsh, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, New Bern, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, North Charleston, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
- Australia (4):
  - Research Site, Nedlands
  - Research Site, South Brisbane
  - Research Site, Spearwood
  - Research Site, Tarragindi
- Canada (5):
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Ajax, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (5):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Písek
  - Research Site, Prague
  - Research Site, Rokycany
- Denmark (5):
  - Research Site, Aalborg
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
- Germany (7):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Darmstadt
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
- Hungary (7):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Edelény
  - Research Site, Gödöllő
  - Research Site, Hajdúnánás
  - Research Site, Pécs
- Israel (3):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Rehovot
- Netherlands (3):
  - Research Site, Eindhoven
  - Research Site, Rotterdam
  - Research Site, Zutphen
- New Zealand (4):
  - Research Site, Auckland
  - Research Site, Christchurch
  - Research Site, Tauranga
  - Research Site, Wellington
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Tarnów
  - Research Site, Wroclaw
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Tygervalley
- Spain (7):
  - Research Site, Alzira
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Mérida
  - Research Site, Salamanca
  - Research Site, Santander
  - Research Site, Zaragoza
- Taiwan (3):
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan
- United Kingdom (5):
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9180C00002&attachmentIdentifier=8cec254d-22b5-4324-a9c7-3a1c85961135&fileName=d9180c00002-study-CSR-synopsis-Redacted.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9180C00002&attachmentIdentifier=e07af4eb-a32b-4902-be1c-366581ef5363&fileName=D9180C00002_-_Statistical_Analysis_Plan-Redacted.pdf&versionIdentifier=
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9180C00002&attachmentIdentifier=0b28d766-11db-42c1-a3d3-a43b0d7d053c&fileName=D9180C00002_-_Protocol_Amendment-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 47 centers in 12 countries (Australia, Canada, Czech Republic, Denmark, Germany, United Kingdom, Hungary, Israel, Poland, South Africa, Spain, and USA).
Pre-assignment Details: A total of 137 participants were randomized, of which 135 participants received at least one dose of study drug.
Period: Overall Study
Arm/Group | Tozorakimab | Placebo
Started | 69 | 68
Treated | 67 | 68
Completed | 58 | 63
Not Completed | 11 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Reason unspecified | 1 | 0
Not completed — Failure to meet randomization criteria | 2 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tozorakimab | Placebo | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (8.3) | 64.3 (6.1) | 64.4 (7.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 41 | 41 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 66 | 66 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 64 | 65 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Pre-bronchodilator Forced Expiratory Volume in 1 Second (Pre-BD FEV1) as Measured in Clinic
Description: The mean change from baseline in Pre-BD FEV1 at Week 12 (tozorakimab - placebo) estimated using a repeated measures mixed effects analysis of covariance measures was estimated. Data available from all visits up to and including Week 12, irrespective of whether the participant discontinued study drug or received reliever therapy was considered. FEV1 was measured by spirometry at clinic.
Time Frame: Baseline (Day -35 to Day -28) through Week 12
Population: Intent-to-treat (ITT) population included all participants who received any study drug and were analyzed according to the treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Litre | 0.019 (0.026) | -0.005 (0.025)
Statistical Analysis 1: Comparison: Tozorakimab vs Placebo; Test type: Other; p = 0.216, Mixed Models Analysis; LS Mean Difference = 0.024, 80% CI 2-sided [-0.015 to 0.063]

2. Secondary Outcome: Serum Tozorakimab Concentration
Description: Serum concentration of tozorakimab collected over time are reported. The lower limit of quantification (LLOQ) for tozorakimab was considered to be 10 μg/L.
Time Frame: Post-dose at Study Weeks 2, 4, 12, 20, 24, 28, 32, and 36
Population: Pharmacokinetic (PK) evaluable population included participants who received at least 1 dose of tozorakimab and had at least 1 detectable post-treatment sample available. Number of participants analyzed (N) denotes the number of participants evaluated for this outcome measure. Number analyzed (n) denotes those participants who had adequate PK sample available at the specified time point.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Tozorakimab
Number analyzed (Participants) | 65
μg/L
  Week 2: number analyzed (Participants) | 64
  Week 2 | 24604.70 (43934.55)
  Week 4 | 8041.59 (22355.66)
  Week 12: number analyzed (Participants) | 63
  Week 12 | 7548.78 (6416.68)
  Week 20: number analyzed (Participants) | 62
  Week 20 | 10789.81 (31903.70)
  Week 24: number analyzed (Participants) | 58
  Week 24 | 6410.05 (4123.46)
  Week 28: number analyzed (Participants) | 58
  Week 28 | 7289.36 (5331.35)
  Week 32: number analyzed (Participants) | 57
  Week 32 | 1483.19 (1779.88)
  Week 36: number analyzed (Participants) | 58
  Week 36 | 420.13 (701.12)

3. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to Tozorakimab
Description: Number of participants with positive ADA to tozorakimab are reported. Treatment-induced ADA positive is defined as ADA negative at baseline and positive at post-baseline assessment. Treatment-boosted ADA positive is defined as ADA positive at baseline and boosted (>= 4 fold) the pre-existing titre during the study period. Persistent positive is defined as ADA negative at baseline and positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or ADA positive at last post-baseline assessment. Transiently positive is defined as ADA negative at baseline and at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: Pre-dose at Study Weeks 0 (baseline) and post-dose at Study Weeks 2, 4, 12, 20, 24, 28, 32, and 36
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who had at least one post-baseline ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 66 | 65
Participants
  Treatment-induced ADA | 1 | 0
  Treatment-boosted ADA | 0 | 0
  Persistently positive ADA | 0 | 0
  Transiently positive ADA | 1 | 0

4. Secondary Outcome: Number of Participants Experiencing First Chronic Obstructive Pulmonary Disease Composite Exacerbations (COPDCompEx) Event
Description: The COPDCompEx combines exacerbations with events defined from participant e-Diaries and peak expiratory flow (PEF). COPDCompEx defined exacerbations included episodes leading to one or more of the following: hospitalization, emergency room visit, treatment with systemic corticosteroids (injected and/or oral), or treatment with antibiotics. Diary COPDCompEx events are defined by threshold and slope criteria being met for >= 2 consecutive days using the following diary and home spirometry variables: overall symptom rating, night-time awakenings due to symptoms, reliever medication use, PEF.
Time Frame: Baseline (Day -35 to Day -28) through Week 28
Population: ITT population included all participants who received any study drug and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants | 28 | 36
Statistical Analysis 1: Comparison: Tozorakimab vs Placebo; Test type: Superiority; p = 0.186, Regression, Cox; Hazard Ratio (HR) = 0.79, 80% CI 2-sided [0.57 to 1.11]

5. Secondary Outcome: Change From Baseline to Week 12 in 4-weekly Mean Evaluating Respiratory Symptoms of COPD (E-RS:COPD) Total Score
Description: Change from baseline to Week 12 in 4-weekly mean E-RS:COPD total score is reported. The E-RS™:COPD is an 11-item electronic patient reported outcome (ePRO) questionnaires developed to evaluate the severity of respiratory symptoms of COPD including breathlessness (5 items; score range: 0 to 17), cough and sputum (3 items; score range: 0 to 11), and chest symptoms (3 items; score range: 0 to 12). The ePRO was completed every day at home and at site visits. Summation of E-RS:COPD item responses produced a total score ranging from 0 to 40, with higher scores indicating greater severity. The 4-weekly mean will be calculated as the sum of all non-missing daily scores over the 28-day evaluation period, divided by the number of non-missing daily scores.
Time Frame: Baseline (from evening of Study Day -14 to the morning of Study Day 1) through Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Units on a scale | -6.09 (1.004) | -6.06 (0.962)

6. Secondary Outcome: Change From Baseline to Week 12 in Mean Breathlessness, Cough and Sputum Scale (BCSS) Score (Over the Previous 4 Weeks)
Description: Change from baseline to Week 12 in mean BCSS score (over the previous 4 weeks) is reported. The BCSS was a 3-item daily diary that assesses the severity of the 3 symptoms: breathlessness, sputum, and cough, each on a 5-point Likert scale ranging from 0 (no symptoms) to 4 (severe symptoms). Item scores were summed to yield a total score ranging from 0 to 12; wherein higher total score indicated more severe symptoms. The BCSS was captured each evening via eDiary. The 4-weekly mean BCSS score was calculated as the sum of all non-missing daily scores over the 28-dayevaluation period, divided by the number of non-missing daily scores.
Time Frame: Baseline (from evening of Study Day -14 to the morning of Study Day 1) through Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Units on a scale | -2.18 (0.313) | -2.18 (0.298)

7. Secondary Outcome: Change From Baseline to Week 12 in Cough Visual Analogue Scale (VAS) Score
Description: Change from baseline to Week 12 in cough VAS score is reported. Participants were asked to complete a cough severity VAS (100 mm linear scale marked with a horizontal line by the participant, with 0 mm representing ''no cough'' and 100 mm representing "worst cough") that measured subjective assessment by the participant of the prior 24 hrs for severity of cough symptoms. It was completed each evening in the eDiary. The 4-weekly mean cough VAS score was calculated as the sum of all non-missing daily scores over the 28-day evaluation period, divided by the number of non-missing daily scores.
Time Frame: Baseline (from evening of Study Day -14 to the morning of Study Day 1) through Week 12
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
mm | -17.21 (3.639) | -17.70 (3.483)

8. Secondary Outcome: Change From Baseline to Week 12 in Saint George's Respiratory Questionnaire (SGRQ) Total Score
Description: Change from baseline to Week 12 in SGRQ total score is reported. The SGRQ was a 50-item electronic PRO instrument developed to measure the health status of participants with airway obstruction diseases and is divided into 2 parts. Part 1 consisted 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; Part 2 consisted 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The SGRQ yielded a total score and three domain scores (symptoms, activity, and impacts). The total score indicated the impact of disease on overall health status, which was expressed as a percentage of overall impairment, in which 100 represents the worst possible health status and 0 indicates the best possible health status. The domain scores range from 0 to 100, with higher scores indicative of greater impairment.
Time Frame: Baseline (from evening of Study Day -14 to the morning of Study Day 1) through Week 12
Population: ITT population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were evaluable at Week 12.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 62 | 64
Units on a scale | -9.177 (2.116) | -8.273 (2.029)

9. Secondary Outcome: Percentage of Participants With a Decrease in SGRQ Total Score of >= 4 Points From Baseline to Week 12
Description: Percentage of participants with a decrease in SGRQ total score of >= 4 points from baseline to Week 12 is reported. The SGRQ was a 50-item electronic PRO instrument developed to measure the health status of participants with airway obstruction diseases and is divided into 2 parts. Part 1 consisted 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; Part 2 consisted 42 items related to the daily activity and psychosocial impacts of individual's respiratory condition. SGRQ yielded a total score and three domain scores (symptoms, activity, and impacts). Total score indicated the impact of disease on overall health status, which was expressed as a percentage of overall impairment, in which 100 represents worst possible health status and 0 indicates best possible health status. The domain scores range from 0 to 100, with higher scores indicative of greater impairment. A change of 4 units/points is associated with a minimum clinically important difference.
Time Frame: Baseline (from evening of Study Day -14 to the morning of Study Day 1) through Week 12
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 62 | 65
Percentage of Participants | 61.3 [0.62 to 1.58] | 61.5

10. Secondary Outcome: Change From Baseline to Week 12 in Airwave Oscillometry (AO) Parameters
Description: Change from baseline to Week 12 in AO parameters including frequency dependence of resistance at 5-20 Hz (R5-R20) and respiratory resistance at 5 Hz (R5; total airway resistance) and 20 Hz (R20; resistance of large airways) is reported. AO is a non-invasive lung function test assessed using an AO device. It is assessed during quiet, tidal breathing with no participant effort required, by superimposing a multi-frequency oscillation onto the participant's natural breathing. AO device uses a vibrating mesh to generate a multifrequency sinusoidal pseudorandom noise (PRN) signal. The AO markers; respiratory resistance at 5 Hz (R5) and 20 Hz (R20) and difference between resistance at 5 and 20Hz (R5-R20; resistance in small airways) are recorded. These markers measure peripheral airway resistance.
Time Frame: Baseline (Study Day 1) and Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: kPa*s/L
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 64 | 66
kPa*s/L
  R5-R20 | 0.008 (0.013) | -0.014 (0.013)
  R5 | 0.015 (0.032) | -0.030 (0.030)
  R20 | 0.006 (0.024) | -0.017 (0.023)

11. Secondary Outcome: Change From Baseline to Week 12 in AO Parameter-Area Under the Reactance Curve (AX)
Description: Change from baseline to Week 12 in AO Parameter-Area Under the Reactance Curve (AX) is reported. AO is a non-invasive lung function test assessed using an AO device. It is assessed during quiet, tidal breathing with no participant effort required, by superimposing a multi-frequency oscillation onto the participant's natural breathing.
Time Frame: Baseline (Study Day 1) and Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: kPa/L
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 64 | 66
kPa/L | -0.081 (0.375) | -0.267 (0.360)

12. Secondary Outcome: Ratio to Baseline in Daily, Night-time, and Awake Time Cough Frequency at Week 12
Description: Ratio to baseline in daily, night-time, and awake time cough frequency at Week 12 is reported. Objective cough frequency was measured using an ambulatory cough monitoring (ACM) which was fitted and worn by the participants for approximately 24 hours after the visits. Daily cough frequency as full average hourly cough of the full duration of recording, night time cough frequency as sleep average hourly cough of the duration of recording at night, and awake time cough frequency as awake average hourly cough of the full duration of recording minus sleep recording will be derived from the recording.
Time Frame: Baseline (Day -21 to Day -7) and Week 12
Population: as for outcome 8
Measure: Geometric Least Squares Mean (80% Confidence Interval); unit: Ratio to baseline
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 58 | 61
Ratio to baseline
  Daily cough frequency | 0.89 [0.74 to 1.07] | 0.83 [0.70 to 0.99]
  Night-time cough frequency | 1.03 [0.62 to 1.70] | 0.61 [0.38 to 0.98]
  Awake time cough frequency | 0.89 [0.74 to 1.07] | 0.84 [0.71 to 0.99]

13. Secondary Outcome: Change From Baseline in Pre-BD FEV1 and Post-BD FEV1 Through Week 28 in Participants With Extent of Emphysema < 10%
Description: Change from baseline in pre-BD FEV1 and post-BD FEV1 through Week 28 in participants with extent of emphysema < 10% is reported.
Time Frame: Baseline (Week -5 to -4) through Week 28 post-dose
Population: ITT population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were evaluable at Week 28.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 31 | 35
Litre
  Pre-BD FEV1 | 0.031 (0.057) | 0.006 (0.049)
  Post-BD FEV1: number analyzed (Participants) | 30 | 34
  Post-BD FEV1 | -0.039 (0.071) | -0.018 (0.059)

14. Secondary Outcome: Change From Baseline in Pre-BD FEV1 and Post-BD FEV1 Through Week 28 in Participants With Extent of Emphysema >= 10%
Description: Change from baseline in pre-BD FEV1 and post-BD FEV1 through Week 28 in participants with extent of emphysema >= 10% is reported.
Time Frame: Baseline (Week -5 to -4) through Week 28 post-dose
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 29 | 29
Litre
  Pre-BD FEV1 Week 28 | -0.015 (0.036) | -0.068 (0.034)
  Post-BD FEV1 Week 28 | 0.074 (0.044) | -0.053 (0.042)

15. Secondary Outcome: Change From Baseline in Pre-BD and Post-BD Forced Vital Capacity (FVC) Through Week 28 in Participants With Extent of Emphysema < 10%
Description: Change from baseline in pre-BD and post-BD FVC through Week 28 in participants with extent of emphysema < 10% is reported.
Time Frame: Baseline (Week -5 to -4) through Week 28 post-dose
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 31 | 35
Litre
  Pre-BD FVC Week 28 | -0.143 (0.105) | -0.056 (0.093)
  Post-BD FVC Week 28: number analyzed (Participants) | 30 | 34
  Post-BD FVC Week 28 | -0.121 (0.114) | 0.046 (0.096)

16. Secondary Outcome: Change From Baseline in Pre-BD and Post-BD FVC Through Week 28 in Participants With Extent of Emphysema >= 10%
Description: Change from baseline in pre-BD and post-BD FVC through Week 28 in participants with extent of emphysema >= 10% is reported.
Time Frame: Baseline (Week -5 to -4) through Week 28 post-dose
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 29 | 29
Litre
  Pre-BD FVC Week 28 | 0.089 (0.086) | -0.121 (0.084)
  Post-BD FVC Week 28 | 0.081 (0.081) | -0.094 (0.077)

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), and TEAEs of Special Interest (TEAESIs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Adverse event of special interest (AESI) are AEs of scientific and medical interest specific to understanding of tozorakimab and requires close monitoring. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 253 days (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants
  Any TEAEs | 53 | 50
  Any TESAEs | 14 | 9
  Any TEAESIs | 33 | 24

18. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (oral or tympanic temperature, diastolic blood pressure, systolic blood pressure, heart [pulse] rate, and respiratory rate).
Time Frame: Day 1 through 253 days (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants
  Hypertension | 2 | 3
  Hypotension | 1 | 0
  Dyspnoea | 2 | 3
  Pyrexia | 1 | 0

19. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of clinical chemistry, hematology, endocrinology, and urinalysis.
Time Frame: Day 1 through 253 days (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants
  Anaemia | 0 | 1
  Hypercholesterolaemia | 0 | 1
  Hyperuricaemia | 0 | 1
  Hypertransaminasaemia | 1 | 0
  Haematuria | 2 | 0
  SARS-CoV-2 test positive | 2 | 0
  Hyperthyroidism | 0 | 1
  Hypothyroidism | 1 | 0
  Urinary tract infection | 0 | 1

20. Secondary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs
Description: Number of participants with abnormal ECGs reported as TEAEs are reported.
Time Frame: Day 1 through 253 days (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants | 1 | 0

21. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) as Measured by Echocardiogram
Description: Change from baseline in LVEF as measured by echocardiogram is reported.
Time Frame: Baseline (Week -3 to -1) through Week 28
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were evaluable at Week 28.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 56 | 60
Ratio | 0.9 (5.78) | 0.2 (4.61)

22. Secondary Outcome: Change From Baseline in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) Level
Description: Change in NT-proBNP Level from baseline is reported.
Time Frame: Baseline (Day -35 to Day -28) through Week 28
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 58 | 61
pmol/L | 4.051 (17.937) | 1.948 (14.280)

23. Secondary Outcome: Number of Participants With Coronavirus Disease 2019 (COVID-19) Related AEs and SAEs
Description: The number of participants with COVID-19 related AEs and SAEs are reported.
Time Frame: Day 1 through 253 days (maximum observed duration)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 67 | 68
Participants
  COVID-19 related AEs | 17 | 14
  COVID-19 related SAEs | 1 | 0

24. Secondary Outcome: Number of Participants Seropositive for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
Description: Number of participants who were seronegative at baseline and who had positive SARS-Cov-2 serology result at the end of study is reported.
Time Frame: Baseline (Week 0) through Week 28
Population: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes the number of participants who were SARS-CoV-2 serum negative at baseline and had at least one post-baseline result.
Measure: Count of Participants; unit: Participants
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 6 | 7
Participants | 6 | 6

25. Other Pre Specified Outcome: Change From Baseline in Post-BD FEV1 To Weeks 12 and 28
Description: Change from baseline in post-BD FEV1 to Weeks 12 and 28 is reported.
Time Frame: Baseline (Week -5 to -4) to Weeks 12 and 28 post-dose
Population: ITT population included all participants who received any study drug and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Litre
Arm/Group | Tozorakimab | Placebo
Number analyzed (Participants) | 65 | 67
Litre
  Week 12 | 0.041 (0.036) | -0.025 (0.033)
  Week 28 | 0.021 (0.036) | -0.049 (0.033)
Statistical Analysis 1: Comparison: Tozorakimab vs Placebo; Results are based on the mixed model for repeated measures (MMRM) analysis at Week 12; Test type: Superiority; p = 0.044, Mixed Models Analysis — One-sided p-value; Kenward-Roger correction has been used for degrees of freedom approximation in the generation of model; Least square mean difference = 0.067, 80% CI 2-sided [0.017 to 0.116]
Statistical Analysis 2: Comparison: Tozorakimab vs Placebo; Results are based on the MMRM analysis at Week 28; Test type: Superiority; p = 0.036, Mixed Models Analysis — One-sided p-value; Kenward-Roger correction has been used for degrees of freedom approximation in the generation of model; Least square mean difference = 0.070, 80% CI 2-sided [0.020 to 0.120]

ADVERSE EVENTS:
Time Frame: Day 1 through 253 days (maximum observed duration)
Description: As-treated population included all participants who received any study drug and were analyzed according to the treatment they actually received.
Arm/Group | Tozorakimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/68
Serious Adverse Events (participants affected / at risk) | 14/67 | 9/68
Other Adverse Events (participants affected / at risk) | 40/67 | 39/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tozorakimab (N=67) | Placebo (N=68)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tozorakimab (N=67) | Placebo (N=68)
Headache (Nervous system disorders) | 8 (10) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 26 (53) | 27 (56)
Injection site erythema (General disorders) | 10 (25) | 0 (0)
Covid-19 (Infections and infestations) | 14 (15) | 14 (14)
Nasopharyngitis (Infections and infestations) | 3 (4) | 7 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04631016/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT04631016/SAP_001.pdf